CLINICAL TRIAL: NCT01695486
Title: Sedation Monitoring During Open Muscle Biopsy in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Eva Tschiedel, MD, University Hospital, Essen
Other Study IDs: 11-4778-BO
Record Dates: First submitted 2012-09-25; First posted 2012-09-28 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Sedation Monitoring in Children
Keywords: BIS; Comfort; open muscle biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare sedation monitoring by bispectral index and comfort score during open muscle biopsies in children.

ELIGIBILITY:
Inclusion Criteria:

* infants, children, adolescents undergoing open muscle biopsy as diagnostic procedure

Exclusion Criteria:

* missing caregiver or patient consent
* intolerance of sedative agents in patients´medical history
* structural brain abnormalities

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children aged 1-18 years undergoing open muscle biopsy as diagnostic procedure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Tschiedel, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Tschiedel E, Muller O, Schara U, Felderhoff-Muser U, Dohna-Schwake C. Sedation monitoring during open muscle biopsy in children by Comfort Score and Bispectral Index - a prospective analysis. Paediatr Anaesth. 2015 Mar;25(3):265-71. doi: 10.1111/pan.12547. Epub 2014 Oct 3. PMID 25279930